CLINICAL TRIAL: NCT06651593
Title: Phase II Biomarker Study of SAR444881 in Combination With Cemiplimab in Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0829; NCI-2024-08852 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with SAR444881 and Cemiplimab (Experimental): SAR444881 will be given by vein over about 60 minutes on Day 1 of each cycle. Cemiplimab will be administered by vein over about 30 minutes on Day 1 of each cycle, starting with Cycle 2. During Cycle 1, you will only receive SAR444881. Starting on Day 1 of Cycle 2 and for all other cycles, you will receive both SAR444881 and cemiplimab.
  Interventions: Drug: SAR444881; Drug: Cemiplimab

INTERVENTIONS:
Drug: SAR444881 — Given by IV
Drug: Cemiplimab — Given by Iv

SUMMARY:
To study possible biomarkers that may be related to how SAR444881 works (either alone or when combined with cemiplimab) in participants with solid tumors.

DETAILED DESCRIPTION:
Primary Objective

* To identify biomarkers:

  * Related to the mechanism of action of SAR444881 alone and in combination with cemiplimab in participants with solid tumors
  * Predictive of response/survival and resistance to the combination of SAR444881 and cemiplimab in participants with solid tumors
* To evaluate the association of biomarkers with response/survival and resistance*:

  * Objective response rate (ORR)
  * Clinical benefit rate (CBR)
  * Progression-free survival (PFS)
  * Overall survival (OS)

Secondary Objectives

* To evaluate the efficacy of the SAR444881 and cemiplimab combination
* To determine the safety and tolerability of the SAR444881 and cemiplimab combination

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an informed consent form (ICF) prior to initiation of the study and any study procedures.
2. Age 18 years.
3. Participants with histologically documented locally advanced or metastatic solid tumor:

   * Cohort 1: NSCLC
   * Cohort 2: MSS CRC and ovarian cancer
4. Prior 10 therapy exposure (Cohort 1 only).
5. Anti-PD-1/PD-L1 na"i"ve (Cohort 2 only).
6. One lesion suitable for repeat biopsy without significant risk to the patient.
7. Measurable disease per the Response Evaluation Criteria in Solid Tumors. Measurable disease should not be the lesion needed for repeat biopsy.
8. Eastern Cooperative Oncology Group (ECOG) performance status of O or 1.
9. Adequate organ and marrow function as defined below within 28 days of study treatment initiation:

   * Hemoglobin >9.0 g/dl (red blood cell/plasma transfusion is not allowed within 2 weeks prior to screening assessment erythropoiesis-stimulating agents/colony- stimulating factors are not allowed within 1 week prior to screening assessment)
   * Absolute neutrophil count 1500/ml (growth factors are not allowed within 2 weeks prior to screening assessment)
   * Platelets 75,000/ml
   * Total bilirubin $1.5 x institutional upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is $3 x ULN.
   * Aspartate transaminase/ALT $2.5 x institutional ULN. Transaminases up to 5 x ULN in the presence of liver metastases.
   * Serum creatinine $1.5 x ULN OR measured or calculated creatinine clearance (CrCI; glomerular filtration rate can also be used in place of creatinine or CrCI) 30 ml/min for patients with creatinine levels >1.5 x institutional ULN (CrCI should be calculated per institutional standard)
   * For participants not receiving therapeutic anticoagulation: international normalized ratio or activated partial thromboplastin time :51.5 x ULN. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
10. Life expectancy 3 months.
11. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result at screening.
12. WOCBP must agree to use adequate contraception for the duration of study participation and for 10 months after completion of study treatment. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a post- menopausal state ( 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Mi..illerian agenesis). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
13. Male participants of childbearing potential must agree to use adequate contraception for the duration of study participation and for 7 months after completion of study treatment. In addition, male participants must be willing to refrain from sperm donation during this time.
14. Willing to undergo mandatory biopsies and blood collections as required by the study.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs.
2. Participants who are pregnant or breastfeeding.
3. Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study treatment initiation. Inhaled or topical steroids, and adrenal replacement steroid doses 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
5. Known history of positive test for human immunodeficiency virus or known acquired immunodeficiency syndrome.
6. Participants with acute hepatitis B virus (HBV) or hepatitis C virus (HCV) infection will be excluded. Participants with chronic HBV or HCV with undetectable viral load will be eligible.
7. Previous solid organ or allogeneic HSCT.
8. Known brain or leptomeningeal metastases.
9. Active infection requiring IV antibiotics or other uncontrolled intercurrent illness requiring hospitalization.
10. Unresolved toxicities from prior therapy (defined as having not resolved to :51 Grade or baseline) or any other toxicity that is deemed irreversible by the investigator. Exceptions include endocrinopathies from prior therapy or disease and successfully treated (such as hypothyroidism, diabetes mellitus), alopecia, vitiligo, and :5 Grade 2 peripheral neuropathy.
11. Participants who have previously been treated with PD-1, PD-L1, or CTLA-4 inhibitors and required permanent discontinuation or systemic immunosuppression due to irAEs (Cohort 1 only).
12. Participants who are receiving any other investigational agents.
13. Treatment with a live, attenuated vaccine within 4 weeks prior to study treatment initiation, or anticipation of need for such a vaccine during the course of the study or within 5 months after the last dose of study treatment.
14. Participants must have adequate washout from prior therapy at the time of study treatment initiation: 4 weeks from major surgery; 4 weeks from antibody-based therapy; 2 weeks or 5 half-lives (whichever is shorter) from any targeted therapy or small molecule therapy; 3 weeks or 5 half-lives (whichever is shorter) from chemotherapy or 6 weeks in the case of certain therapies (e.g., extensive radiotherapy, mitomycin C, and nitrosoureas); and 4 weeks from radiation therapy. Palliative radiotherapy is permitted for a preexisting lesion, provided it does not interfere with the assessment of tumor target lesions (e.g., the lesion to be irradiated must not be a site of measurable disease).
15. Prior treatment with ILT2 or ILT4 inhibitor.
16. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
17. Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
18. Inability to comply with the study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, Md, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Md Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org